CLINICAL TRIAL: NCT01192204
Title: Clinical Evaluation of Bioadhesive Gels for Oral Cancer Chemoprevention
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: University of Louisville (Other); University of North Carolina, Chapel Hill (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan Mallery DDS, PhD, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2009C0086; RC2CA148099 (NIH)
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Results first posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2013-11

CONDITIONS: Squamous Cell Carcinoma of Mouth; Intraepithelial Neoplasia
Keywords: FBR, OSCC, chemoprevention
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma in Situ

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% FBR containing bioadhesive gel (Active Comparator): Drug consisting of 10% FBR containing bioadhesive gel. Participants instructed to apply 0.5 gm of 10% FBR containing bioadhesive gel four times a day to lesional site
  Interventions: Drug: 10% FBR containing bioadhesive gel
- Placebo Gel (Placebo Comparator): Color/consistency matched placebo (no black raspberry) gel
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: 10% FBR containing bioadhesive gel — 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
  Other Names: BRB gel
  Arms: 10% FBR containing bioadhesive gel
Drug: placebo gel — 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
  Other Names: BRB devoid placebo gel
  Arms: Placebo Gel

SUMMARY:
This is a multicenter placebo-controlled clinical trial to assess the effects of a topically applied gel on precancerous oral epithelial lesions. A total of 41 participants will be enrolled in this trial, and 22 of them will be enrolled at Ohio State. [The remaining 19 participants will be enrolled at the University of North Carolina (9 participants) and the University of Louisville (8 participants)]. At all three institutions, half of the participants will randomly be assigned to the 10% FBR gel (0.5 gm four times daily for 3 months), while half will enter the placebo control arm. All trial participants will have a pretreatment (including lesional and perilesional tissue) biopsy taken before and an excisional biopsy after 3 months of treatment. As pretreatment indices are compared to post treatment effects on each patient, patients serve as their own internal control. Pretreatment lesional biopsies are obtained to establish a pretreatment diagnosis and provide a pretreatment baseline for the experimental parameters.

DETAILED DESCRIPTION:
Forty one (41) patients with microscopically confirmed premalignant oral epithelial disease (epithelial dysplasia) will be enrolled in this trial at three clinical centers, i.e. the Ohio State University, University of North Carolina at Chapel Hill and University of Louisville. At all three institutions, half of the participants will randomly be assigned to the 10% FBR gel (0.5 gm four times daily for 3 months), while half will enter the placebo control arm.

In accordance with the established standard of care, all participants need to have biopsies taken of their suspicious oral lesions to establish the diagnosis (non research). Trial participants will have three total biopsies. Pretreatment biopsies will entail: 1) perilesional tissue and single saliva sample for FBR metabolic profiling studies (tissue and saliva will be obtained 15 minutes after a single 0.5 gm application of 10% FBR gel for metabolic profiling. Gel application and nonlesional biopsy will be obtained before incisional biopsy of lesional tissue), and 2) a hemisection of lesional tissue to establish a diagnosis and provide a pretreatment baseline for the experimental parameters. While the pretreatment biopsy includes removal of both perilesional and lesional tissue, there will only be one surgical wound as the perilesional tissue is contiguous with the lesional tissue. A final excisional biopsy of the treatment site including any remaining residual lesional tissue (excision of oral dysplastic lesions is consistent with current standards of care) will be obtained after 3 months of treatment. The experimental design permits each patient to serve as their own internal control. Briefly, these following parameters will be monitored in all participants (comparisons made relative to patient-matched pretreatment to posttreatment biopsies): 1) light microscopic diagnoses, 2) clinical appearances and lesional sizes, 3) microarray gene expression analyses, 4) microvascular densities of superficial connective tissues, 5) LOH indices at loci associated with tumor suppressor genes, 6) intraepithelial levels of COX-2 and iNOS protein (image analysis quantified immunohistochemistry), 7) comparison of FBR metabolic profiles relative to extent of chemopreventive efficacy noted.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 21 to 80
2. Microscopically confirmed premalignant oral epithelial disease
3. No previous history of cancer (with the exception of basal cell carcinoma of the skin)
4. Tobacco free for at least six weeks prior to entrance in the trial and remain tobacco-free for the three month duration of the study
5. Availability for necessary study follow-up evaluations (every 10 to 14 days during the trial)
6. Capable of providing informed consent.

Exclusion Criteria:

1. Previous history of cancer (with the exception of basal cell carcinoma of the skin)
2. Current use of tobacco products or refusal to remain tobacco-free for the three month duration of the study
3. Lack of microscopically confirmed premalignant oral epithelial changes
4. Microscopic diagnosis of oral squamous cell carcinoma
5. Previous history of radiation therapy on same side of the head and neck region
6. History of allergy to any kind of berry
7. Women who are determined to be pregnant or plan to be pregnant during the trial
8. Women who are nursing.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan R Mallery, DDS, PhD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - University of Louisville, School of Dentistry, Louisville, Kentucky
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - The Ohio State University, College of Dentistry, Columbus, Ohio

REFERENCES:
- [Background] Menzin J, Lines LM, Manning LN. The economics of squamous cell carcinoma of the head and neck. Curr Opin Otolaryngol Head Neck Surg. 2007 Apr;15(2):68-73. doi: 10.1097/MOO.0b013e328017f669. PMID 17413405
- [Background] Lefebvre JL. Current clinical outcomes demand new treatment options for SCCHN. Ann Oncol. 2005;16 Suppl 6:vi7-vi12. doi: 10.1093/annonc/mdi452. PMID 15987995
- [Background] Papadimitrakopoulou VA, Clayman GL, Shin DM, Myers JN, Gillenwater AM, Goepfert H, El-Naggar AK, Lewin JS, Lippman SM, Hong WK. Biochemoprevention for dysplastic lesions of the upper aerodigestive tract. Arch Otolaryngol Head Neck Surg. 1999 Oct;125(10):1083-9. doi: 10.1001/archotol.125.10.1083. PMID 10522499
- [Background] Rudin CM, Cohen EE, Papadimitrakopoulou VA, Silverman S Jr, Recant W, El-Naggar AK, Stenson K, Lippman SM, Hong WK, Vokes EE. An attenuated adenovirus, ONYX-015, as mouthwash therapy for premalignant oral dysplasia. J Clin Oncol. 2003 Dec 15;21(24):4546-52. doi: 10.1200/JCO.2003.03.544. Epub 2003 Nov 3. PMID 14597742
- [Background] Lippman SM, Lee JJ, Martin JW, El-Naggar AK, Xu X, Shin DM, Thomas M, Mao L, Fritsche HA Jr, Zhou X, Papadimitrakopoulou V, Khuri FR, Tran H, Clayman GL, Hittelman WN, Hong WK, Lotan R. Fenretinide activity in retinoid-resistant oral leukoplakia. Clin Cancer Res. 2006 May 15;12(10):3109-14. doi: 10.1158/1078-0432.CCR-05-2636. PMID 16707609
- [Background] Toma S, Benso S, Albanese E, Palumbo R, Cantoni E, Nicolo G, Mangiante P. Treatment of oral leukoplakia with beta-carotene. Oncology. 1992;49(2):77-81. doi: 10.1159/000227016. PMID 1574255
- [Background] Lippman SM, Batsakis JG, Toth BB, Weber RS, Lee JJ, Martin JW, Hays GL, Goepfert H, Hong WK. Comparison of low-dose isotretinoin with beta carotene to prevent oral carcinogenesis. N Engl J Med. 1993 Jan 7;328(1):15-20. doi: 10.1056/NEJM199301073280103. PMID 8416267
- [Background] Shin DM, Mao L, Papadimitrakopoulou VM, Clayman G, El-Naggar A, Shin HJ, Lee JJ, Lee JS, Gillenwater A, Myers J, Lippman SM, Hittelman WN, Hong WK. Biochemopreventive therapy for patients with premalignant lesions of the head and neck and p53 gene expression. J Natl Cancer Inst. 2000 Jan 5;92(1):69-73. doi: 10.1093/jnci/92.1.69. No abstract available. PMID 10620636
- [Background] Papadimitrakopoulou VA, William WN Jr, Dannenberg AJ, Lippman SM, Lee JJ, Ondrey FG, Peterson DE, Feng L, Atwell A, El-Naggar AK, Nathan CO, Helman JI, Du B, Yueh B, Boyle JO. Pilot randomized phase II study of celecoxib in oral premalignant lesions. Clin Cancer Res. 2008 Apr 1;14(7):2095-101. doi: 10.1158/1078-0432.CCR-07-4024. PMID 18381950
- [Background] William WN Jr, Lee JJ, Lippman SM, Martin JW, Chakravarti N, Tran HT, Sabichi AL, Kim ES, Feng L, Lotan R, Papadimitrakopoulou VA. High-dose fenretinide in oral leukoplakia. Cancer Prev Res (Phila). 2009 Jan;2(1):22-6. doi: 10.1158/1940-6207.CAPR-08-0100. PMID 19139014
- [Background] Meyskens FL Jr. Another negative chemoprevention trial: what can we learn? Clin Cancer Res. 2008 Jan 1;14(1):2-3. doi: 10.1158/1078-0432.CCR-07-2215. No abstract available. PMID 18172244
- [Background] Rodrigo KA, Rawal Y, Renner RJ, Schwartz SJ, Tian Q, Larsen PE, Mallery SR. Suppression of the tumorigenic phenotype in human oral squamous cell carcinoma cells by an ethanol extract derived from freeze-dried black raspberries. Nutr Cancer. 2006;54(1):58-68. doi: 10.1207/s15327914nc5401_7. PMID 16800773
- [Background] Chen T, Rose ME, Hwang H, Nines RG, Stoner GD. Black raspberries inhibit N-nitrosomethylbenzylamine (NMBA)-induced angiogenesis in rat esophagus parallel to the suppression of COX-2 and iNOS. Carcinogenesis. 2006 Nov;27(11):2301-7. doi: 10.1093/carcin/bgl109. Epub 2006 Jun 15. PMID 16777990
- [Background] Chen T, Hwang H, Rose ME, Nines RG, Stoner GD. Chemopreventive properties of black raspberries in N-nitrosomethylbenzylamine-induced rat esophageal tumorigenesis: down-regulation of cyclooxygenase-2, inducible nitric oxide synthase, and c-Jun. Cancer Res. 2006 Mar 1;66(5):2853-9. doi: 10.1158/0008-5472.CAN-05-3279. PMID 16510608
- [Background] Kresty LA, Morse MA, Morgan C, Carlton PS, Lu J, Gupta A, Blackwood M, Stoner GD. Chemoprevention of esophageal tumorigenesis by dietary administration of lyophilized black raspberries. Cancer Res. 2001 Aug 15;61(16):6112-9. PMID 11507061
- [Background] Xue H, Aziz RM, Sun N, Cassady JM, Kamendulis LM, Xu Y, Stoner GD, Klaunig JE. Inhibition of cellular transformation by berry extracts. Carcinogenesis. 2001 Feb;22(2):351-6. doi: 10.1093/carcin/22.2.351. PMID 11181460
- [Background] Huang C, Huang Y, Li J, Hu W, Aziz R, Tang MS, Sun N, Cassady J, Stoner GD. Inhibition of benzo(a)pyrene diol-epoxide-induced transactivation of activated protein 1 and nuclear factor kappaB by black raspberry extracts. Cancer Res. 2002 Dec 1;62(23):6857-63. PMID 12460899
- [Background] Huang C, Li J, Song L, Zhang D, Tong Q, Ding M, Bowman L, Aziz R, Stoner GD. Black raspberry extracts inhibit benzo(a)pyrene diol-epoxide-induced activator protein 1 activation and VEGF transcription by targeting the phosphotidylinositol 3-kinase/Akt pathway. Cancer Res. 2006 Jan 1;66(1):581-7. doi: 10.1158/0008-5472.CAN-05-1951. PMID 16397275
- [Background] Hecht SS, Huang C, Stoner GD, Li J, Kenney PM, Sturla SJ, Carmella SG. Identification of cyanidin glycosides as constituents of freeze-dried black raspberries which inhibit anti-benzo[a]pyrene-7,8-diol-9,10-epoxide induced NFkappaB and AP-1 activity. Carcinogenesis. 2006 Aug;27(8):1617-26. doi: 10.1093/carcin/bgi366. Epub 2006 Mar 7. PMID 16522666
- [Background] Stoner GD. Foodstuffs for preventing cancer: the preclinical and clinical development of berries. Cancer Prev Res (Phila). 2009 Mar;2(3):187-94. doi: 10.1158/1940-6207.CAPR-08-0226. Epub 2009 Mar 3. PMID 19258544
- [Background] Wang LS, Hecht SS, Carmella SG, Yu N, Larue B, Henry C, McIntyre C, Rocha C, Lechner JF, Stoner GD. Anthocyanins in black raspberries prevent esophageal tumors in rats. Cancer Prev Res (Phila). 2009 Jan;2(1):84-93. doi: 10.1158/1940-6207.CAPR-08-0155. PMID 19139022
- [Background] Shumway BS, Kresty LA, Larsen PE, Zwick JC, Lu B, Fields HW, Mumper RJ, Stoner GD, Mallery SR. Effects of a topically applied bioadhesive berry gel on loss of heterozygosity indices in premalignant oral lesions. Clin Cancer Res. 2008 Apr 15;14(8):2421-30. doi: 10.1158/1078-0432.CCR-07-4096. PMID 18413833
- [Background] Mallery SR, Zwick JC, Pei P, Tong M, Larsen PE, Shumway BS, Lu B, Fields HW, Mumper RJ, Stoner GD. Topical application of a bioadhesive black raspberry gel modulates gene expression and reduces cyclooxygenase 2 protein in human premalignant oral lesions. Cancer Res. 2008 Jun 15;68(12):4945-57. doi: 10.1158/0008-5472.CAN-08-0568. PMID 18559542
- [Background] Ugalde CM, Liu Z, Ren C, Chan KK, Rodrigo KA, Ling Y, Larsen PE, Chacon GE, Stoner GD, Mumper RJ, Fields HW, Mallery SR. Distribution of anthocyanins delivered from a bioadhesive black raspberry gel following topical intraoral application in normal healthy volunteers. Pharm Res. 2009 Apr;26(4):977-86. doi: 10.1007/s11095-008-9806-x. Epub 2009 Jan 10. PMID 19137418
- [Background] Lang K, Menzin J, Earle CC, Jacobson J, Hsu MA. The economic cost of squamous cell cancer of the head and neck: findings from linked SEER-Medicare data. Arch Otolaryngol Head Neck Surg. 2004 Nov;130(11):1269-75. doi: 10.1001/archotol.130.11.1269. PMID 15545580
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Silverman S Jr, Gorsky M, Lozada F. Oral leukoplakia and malignant transformation. A follow-up study of 257 patients. Cancer. 1984 Feb 1;53(3):563-8. doi: 10.1002/1097-0142(19840201)53:33.0.co;2-f. PMID 6537892
- [Background] Sciubba JJ. Oral leukoplakia. Crit Rev Oral Biol Med. 1995;6(2):147-60. doi: 10.1177/10454411950060020401. PMID 7548621
- [Background] Speight PM. Update on oral epithelial dysplasia and progression to cancer. Head Neck Pathol. 2007 Sep;1(1):61-6. doi: 10.1007/s12105-007-0014-5. Epub 2007 Nov 30. No abstract available. PMID 20614284
- [Background] Helzer LJ, Heitkamp KM, Shein M, Etzel RA. Pilot study of methods to measure saliva cotinine in Alaska Native women during pregnancy. Int J Circumpolar Health. 2007;66 Suppl 1:29-38. PMID 18154230
- [Background] Mao L, Lee JS, Fan YH, Ro JY, Batsakis JG, Lippman S, Hittelman W, Hong WK. Frequent microsatellite alterations at chromosomes 9p21 and 3p14 in oral premalignant lesions and their value in cancer risk assessment. Nat Med. 1996 Jun;2(6):682-5. doi: 10.1038/nm0696-682. PMID 8640560
- [Background] Chan G, Boyle JO, Yang EK, Zhang F, Sacks PG, Shah JP, Edelstein D, Soslow RA, Koki AT, Woerner BM, Masferrer JL, Dannenberg AJ. Cyclooxygenase-2 expression is up-regulated in squamous cell carcinoma of the head and neck. Cancer Res. 1999 Mar 1;59(5):991-4. PMID 10070952
- [Background] Connelly ST, Macabeo-Ong M, Dekker N, Jordan RC, Schmidt BL. Increased nitric oxide levels and iNOS over-expression in oral squamous cell carcinoma. Oral Oncol. 2005 Mar;41(3):261-7. doi: 10.1016/j.oraloncology.2004.09.007. PMID 15743688
- [Background] Kawanishi S, Hiraku Y, Pinlaor S, Ma N. Oxidative and nitrative DNA damage in animals and patients with inflammatory diseases in relation to inflammation-related carcinogenesis. Biol Chem. 2006 Apr;387(4):365-72. doi: 10.1515/BC.2006.049. PMID 16606333
- [Background] Mann JR, Backlund MG, DuBois RN. Mechanisms of disease: Inflammatory mediators and cancer prevention. Nat Clin Pract Oncol. 2005 Apr;2(4):202-10. doi: 10.1038/ncponc0140. PMID 16264935
- [Background] Joshi N, Johnson LL, Wei WQ, Abnet CC, Dong ZW, Taylor PR, Limburg PJ, Dawsey SM, Hawk ET, Qiao YL, Kirsch IR. Gene expression differences in normal esophageal mucosa associated with regression and progression of mild and moderate squamous dysplasia in a high-risk Chinese population. Cancer Res. 2006 Jul 1;66(13):6851-60. doi: 10.1158/0008-5472.CAN-06-0662. PMID 16818663
- [Background] Otrock ZK, Mahfouz RA, Makarem JA, Shamseddine AI. Understanding the biology of angiogenesis: review of the most important molecular mechanisms. Blood Cells Mol Dis. 2007 Sep-Oct;39(2):212-20. doi: 10.1016/j.bcmd.2007.04.001. Epub 2007 Jun 6. PMID 17553709
- [Background] Tong M, Lloyd B, Pei P, Mallery SR. Human head and neck squamous cell carcinoma cells are both targets and effectors for the angiogenic cytokine, VEGF. J Cell Biochem. 2008 Dec 1;105(5):1202-10. doi: 10.1002/jcb.21920. PMID 18802921
- [Background] Kannan R, Bijur GN, Mallery SR, Beck FM, Sabourin CL, Jewell SD, Schuller DE, Stoner GD. Transforming growth factor-alpha overexpression in proliferative verrucous leukoplakia and oral squamous cell carcinoma: an immunohistochemical study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1996 Jul;82(1):69-74. doi: 10.1016/s1079-2104(96)80379-9. PMID 8843456
- [Background] Wang LS, Stoner GD. Anthocyanins and their role in cancer prevention. Cancer Lett. 2008 Oct 8;269(2):281-90. doi: 10.1016/j.canlet.2008.05.020. Epub 2008 Jun 20. PMID 18571839
- [Result] Mallery SR, Tong M, Shumway BS, Curran AE, Larsen PE, Ness GM, Kennedy KS, Blakey GH, Kushner GM, Vickers AM, Han B, Pei P, Stoner GD. Topical application of a mucoadhesive freeze-dried black raspberry gel induces clinical and histologic regression and reduces loss of heterozygosity events in premalignant oral intraepithelial lesions: results from a multicentered, placebo-controlled clinical trial. Clin Cancer Res. 2014 Apr 1;20(7):1910-24. doi: 10.1158/1078-0432.CCR-13-3159. Epub 2014 Jan 31. PMID 24486592

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 41 patients were enrolled in this protocol. 1 patient could not keep the appointments and was referred to his private oral surgeon.
Groups:
- 10% FBR Gel: Active 10% FBR containing bioadhesive gel
  Bioadhesive 10% freeze-dried black raspberry gel: 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
- Placebo Gel: Color/consistency matched placebo (no black raspberry) gel
  Color/consistency matched placebo gel: 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
Period: Overall Study
Arm/Group | 10% FBR Gel | Placebo Gel
Started | 23 | 18
Completed | 22 | 18
Not Completed | 1 | 0
Not completed — could not keep recall appointments | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10% FBR Gel | Placebo Gel | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Categorical [Count of Participants; unit: Participants] — The patients were randomly assigned by computer generated numbers to either the BRB or the placebo gel groups.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 5 | 22
    >=65 years | 6 | 13 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (1.8) | 57.7 (2.9) | 59.9 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 9 | 23
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: Light Microscopic Histologically Scored Diagnoses Pretreatment to Post Treatment
Description: A hemisection of lesional tissue will be conducted before the 3 month treatment to establish a diagnosis and provide a pretreatment baseline for the experimental parameters. Anl excisional biopsy of the treatment site including any remaining residual lesional tissue (excision of oral dysplastic lesions is consistent with current standards of care) will be obtained after 3 months of treatment to provide a posttreatment diagnosis. The 0 to 8 histologic scale was:0=normal with or without hyperkeratosis BEST OUTCOME, 1=atypia, 2=mild dysplasia, 3=mild-moderate dysplasia, 4=moderate dysplasia,5=moderate-severe dysplasia,6=severe dysplasia, 7=carcinoma in situ, 8=invasive oral squamous cell carcinoma (WORST OUTCOME).
Time Frame: Before and after the 3 month treatment.
Population: The population evaluated were as previously described i.e. 22 participants in the BRB gel cohort and 18 participants in the placebo gel cohort.
Measure: Mean (Standard Error); unit: unit on histologic grade scale
Arm/Group | 10% FBR Gel | Placebo Gel
Number analyzed (Participants) | 22 | 18
unit on histologic grade scale
  Pretreatment | 2.36 (0.35) | 2.83 (0.34)
  Posttreatment | 1.9 (0.21) | 2.58 (0.17)
Statistical Analysis 1: Comparison: 10% FBR Gel; Wilcoxon matched-pairs signed rank test (intrapatient pre versus post treatment scores); Test type: Superiority or Other; p = 0.048, Wilcoxon matched-pairs signed rank test — Statistical analyses reflect percent change intrapatient pre versus post histologic grade scores; We used a 2-tailed Mann Whitney U test to evaluate these data
Statistical Analysis 2: Comparison: Placebo Gel; Wilcoxon matched-pairs signed rank test (pre versus post treatment scores); Test type: Superiority or Other; p = 0.50, Wilcoxon matched-pairs signed rank test — Statistical analyses reflect percent change pre versus post histologic grade scores

2. Secondary Outcome: Changes in Lesional Sizes
Description: The remaining oral dysplasia lesion will be inspected at each follow up appointment (every 10-14 days). Biopsies will be immediately conducted on patients with any indication of malignant transformation including indurated, rolled borders, nonhealing ulcers, etc. Accordingly, these patients will withdraw from the trial. Participants will also be monitored for any changes consistent with contact mucositis e.g. soreness and erythema at application site. Clinical photographs were taken for the patients records. Pre treatment and post treatment photographs, with a ruler in place, were used for accurate pre and post treatment size measurement. NOTE: if treatment is beneficial, lesional size will decrease which will be reflected as a negative number.
Time Frame: pretreatment and posttreatment (3 months treatment duration)
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | 10% FBR Gel | Placebo Gel
Number analyzed (Participants) | 22 | 18
mm^2 | -26.12 (5.81) | 18.12 (4.39)
Statistical Analysis 1: Comparison: 10% FBR Gel; Test type: Superiority or Other; p < 0.002, Wilcoxon matched-pairs signed rank test; specifically, we used the Wilcoxon matched-pairs signed rank test
Statistical Analysis 2: Comparison: Placebo Gel; Test type: Superiority or Other; p = 0.036, Wilcoxon matched-pairs signed rank test

3. Secondary Outcome: Treatment Changes in Loss of Heterozygosity Events
Description: Laboratory experiments will be conducted to assess the effects of gel treatment on pre and post loss of heterozygosity (LOH) events at loci associated with tumor suppressor genes.
Time Frame: Before and after the 3 month treatment duration
Measure: Mean (Standard Error); unit: LOH events
Arm/Group | 10% FBR Gel | Placebo Gel
Number analyzed (Participants) | 22 | 18
LOH events | 0.9 (0.02) | 0.4 (0.03)
Statistical Analysis 1: Comparison: 10% FBR Gel; Test type: Superiority or Other; p = 0.002, 2-tailed unpaired t test
Statistical Analysis 2: Comparison: Placebo Gel; Test type: Superiority or Other; p = 0.16, two-tailed unpaired t test

ADVERSE EVENTS:
Groups:
- 10% FBR Gel: Active 10% FBR containing bioadhesive gel
  Bioadhesive 10% freeze-dried black raspberry gel: 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
  No adverse events
- Placebo Gel: Color/consistency matched placebo (no black raspberry) gel
  Color/consistency matched placebo gel: 0.5 gm applied 4 times daily to the oral premalignant lesion site for a duration of 3 months
  No adverse events
Arm/Group | 10% FBR Gel | Placebo Gel
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/22 | 0/18

LIMITATIONS AND CAVEATS:
While we initially planned to include microvascular densities and COX-2 analyses, there were insufficient tissue samples to collect these data. Therefore as we do not have these data we can not report them.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No